CLINICAL TRIAL: NCT01275963
Title: New Echocardiographic Parameters for Assessment of Longitudinal Left Ventricular Function
Acronym: LAX
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Derliz Mereles, Dr. Derliz Mereles, Heidelberg University
Other Study IDs: S-401/2010
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Cardiovascular Pathology
Keywords: Echocardiography; Strain imaging; Ventricular Dysfunction; Cardiomyopathy; Longitudinal left ventricular function
MeSH Terms: conditions — Ventricular Dysfunction; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Control: Healthy individuals without structural heart disease
- CAD: Patients with coronary artery disease
- DCM: Participants with dilated cardiomyopathy
- HNCM: Patients with hypertrophic non-obstructive cardiomyopathy
- HOCM: Patients with hypertrophic obstructive cardiomyopathy
- RCM: Patients with restrictive cardiomyopathy
- Amyloidosis: Patients with cardiac manifestation of amyloidosis
- HFPEF: Patients with heart failure with preserved ejection fraction (diastolic heart failure)

SUMMARY:
Assessment of left ventricular systolic function is the most frequent indication for routine echocardiography. Qualitative eyeball method and biplane modified Simpson's rule, both measuring radial ventricular function, are the currently recommended methods to meet this challenge. Due to the complexity of the myocardial architecture, global left ventricular function also has longitudinal and torsional components.

The aim of this study is to evaluate new echocardiographic parameters for longitudinal left ventricular function. A special focus is set on strain imaging by speckle tracking, which is a relatively new technique. Patients with different cardiac pathologies (e. g. dilated cardiomyopathy, coronary artery disease, diastolic dysfunction) will be included and compared to healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* persons of 18 years and older who receive a transthoracic echocardiography at our department
* written consent

Exclusion Criteria:

* permanent pacemaker rhythm
* moderate/severe valvular heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals and patients with various cardiac pathologies, who undergo routine echocardiography at our department
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
left ventricular longitudinal systolic strain (LV-LSS) in all patients | 2 years
  left ventricular longitudinal systolic strain (LV-LSS) is measured in all patients by speckle tracking strain imaging

SECONDARY OUTCOMES:
mitral annular plane systolic excursion (MAPSE) in all patients | 2 years
  MAPSE is measured by M-Mode echocardiography
mitral annular systolic velocity (MASV) in all patients | 2 years
  MASV is derived from tissue doppler
diastolic left ventricular function in all patients | 2 years
  Diastolic function is assesed by mitral inflow, mitral annulus velocity, pulmonary vein flow and velocity of flow progression.
pulmonary artery systolic pressure (PASP) in all patients | 2 years
  PASP is derived from Tricuspid valve regurgitation velocity
left ventricular ejection fraction (LVEF) in all patients | 2 years
  EF is measured by modified Simpson's rule (biplane)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Aurich, M.D., Principal Investigator — Heidelberg University; Derliz Mereles, M.D., Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Aurich M, Keller M, Greiner S, Steen H, Aus dem Siepen F, Riffel J, Katus HA, Buss SJ, Mereles D. Left ventricular mechanics assessed by two-dimensional echocardiography and cardiac magnetic resonance imaging: comparison of high-resolution speckle tracking and feature tracking. Eur Heart J Cardiovasc Imaging. 2016 Dec;17(12):1370-1378. doi: 10.1093/ehjci/jew042. Epub 2016 Mar 24. PMID 27013249